CLINICAL TRIAL: NCT06757478
Title: A Clinical Study on the Combination of Mitoxantrone Liposome Injection, Bendamustine, Etoposide, and Cytarabine for Pretreatment of Autologous Hematopoietic Stem Cell Transplantation in Patients with Lymphoma
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Principal Investigator, Lixia Sheng, Doctor, First Affiliated Hospital of Ningbo University
Other Study IDs: 2024-157A-01
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma Patient
Keywords: Mitoxantrone hydrochloride liposome; bendamustine; etoposide; cytarabine; HSCT; lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — In this study, the following biological samples were collected: blood samples were collected 10 mL/ time *3 times for each patient, which were used for blood routine, blood biochemistry, cTnI or cTnT, BNP or pro BNP, and infectious disease markers; Urine samples 10mL/ time *3 times for each patient for urine routine detection, women of childbearing age need to collect another 10 ml/time *1 urine sample for pregnancy detection; Bone marrow samples should be collected 8 mL/ time *2 times for bone marrow examination in patients suspected of having bone marrow infiltration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- lymphoma patient: Preconditioning for auto-HSCT

SUMMARY:
This is a single-arm, open, single-center clinical study. Patients with lymphoma who were to undergo autologous hematopoietic stem cell transplantation were pretreated with mitoxantrone hydrochloride liposome injection combined with standard doses of bendamustine, etoposide, and cytarabine before transplantation, in order to explore the safety and efficacy of this combined pretreatment regimen.

Tests were performed during the study to observe efficacy, safety, and tolerability. The treatment period was from pre-treatment to +28 days after transplantation and +28 days after stem cells were transfused. The follow-up period was followed up once a month for 6 months, every 3 months for 6 months to 2 years, and every 6 months for 2 years to 3 years after stem cell reinfusion. All subjects underwent protocol-mandated examinations during treatment to observe safety, tolerability, and efficacy.

DETAILED DESCRIPTION:
In the treatment of malignant lymphoma (ML), autologous hematopoietic stem cell transplantation (ASCT) is one of the important means, and high-dose chemotherapy combined with ASCT is considered to be the standard treatment for chemotherapy sensitive relapsed/refractory (R/R) non-Hodgkin lymphoma (NHL) patients [1,2]. Preconditioning is an important part of ASCT, which refers to high-dose chemotherapy and (or) radiotherapy and immunosuppressive treatment before hematopoietic stem cell transfusion to clear tumor cells in patients and prepare for hematopoietic stem cell transfusion [3]. With the development in recent decades, the preconditioning regimen has also undergone diversified changes. From the whole body irradiation (TBI)/cyclophosphamide (Cy) in the 1970s to the Mafran /Cy in the 1980s [4], various transplant centers have been trying various improved programs. The overall survival rate of different high-dose regimens combined with AHSCT is about 30-70% [5].

The simple chemotherapy transplantation preconditioning regimen without TBI can be divided into camustine (BCNU) and BU-based regimen. BCNU is one of the commonly used alkylating agents and is often combined with VP-16, Arc-C, Cy, Bu to form BEAM, CBV, BEAC and other transplantation preconditioning regimen. BEAM and CBV are the most commonly used solutions. The 5-year OS and 5-year PFS in the treatment of relapsed refractory lymphoma by ASCT with BEAM preconditioning regimen were 44%-71% and 35%-50% [6,7]. Compared with CBV, BuCy, and TBI, BEAM preconditioning showed better survival benefits in 3-year PFS and OS in non-Hodgkin lymphoma autologous transplantation [8].

Due to the high incidence of interstitial pneumonia in lymphoma patients who received a pre-treatment regimen containing high-dose carmostine, a BeEAM regimen (bendamustine, etoposide, cytarabine, mephalam) was replaced with carmostine to reduce toxicity and improve efficacy. Redondo AM et al. [9] reported the results of BeEAM protocol in DLBCL and peripheral T-cell lymphoma in a phase 2 clinical trial: the 3-year PFS and OS were 58% and 75%, respectively, the non-recurrent mortality was similar to that of previous pretreatment regimen, and the incidence of other toxics was lower. Therefore, BeEAM regimen may be a preconditioning regimen that can improve efficacy and reduce toxicity in patients with aggressive NHL. Although BeEAM regimen reduced the incidence of interstitial pneumonia caused by camustine, the adverse reaction caused by mafaran, myelosuppression, was dose-limited toxicity, mainly manifested as leukopenia, thrombocytopenia and anemia, followed by gastrointestinal reactions, including nausea and vomiting. In order to further improve the safety of BeEAM regimen, drugs with similar mechanism and less toxic side effects can be used to replace Mafaran to form a new pretreatment regimen.

Mitoxantrone (MTO) is an anthraquinone antibiotic antitumor agent. Its main mechanism of action is to insert deoxyribonucleic acid through hydrogen bonding, which causes the cross-linking and breaking of DNA structure. Can interfere with RNA; As a topoisomerase II inhibitor, mitoxantrone is a cell cycle non-specific drug that can kill both proliferative and non-proliferative cancer cells in humans [10]. Mitoxantrone injection was used in combination with cyclophosphamide, carazine, and podoside as a preconditioning regimen for autologous peripheral blood stem cell transplantation in a patient with recurrent and refractory Hodgkin's disease, and the transplantation was successful with only mild gastrointestinal reaction. Mitoxantrone injection and Mafaran combined to compare the application effect of BEAM in ASCT preconditioning of lymphoma patients, the results showed that the OS of the two groups was similar, and the PFS of CR patients showed no statistical difference between the two groups. Mitoxantrone injection was also compared with the Cy-fTBI regimen combined with bixiaoan and Mafaran when exploring the transplantation preconditioning regimen for patients with non-Hodgkin's lymphoma. There was no statistical difference in remission rate, DFS and OS indexes between the two groups. Mitoxantrone injection combined with bioxan and mafaran significantly improved transplant-related mortality.

The development of mitoxantrone into liposomes to improve the release and distribution of drugs and reduce the side effects of drugs is worthy of the application of mitoxantrone hydrochloride liposomes in the pretreatment of lymphoma patients for autologous transplantation based on the factors of evidence-based medicine, diagnosis and treatment norms, and taking into account the cost-benefit ratio. The purpose of this study was to evaluate the safety and efficacy of mitoxantrone hydrochloride liposome injection combined with bendamustine, etoposide and cytarabine in patients pretreated for lymphoma autologous hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patients voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with the follow-up; 2. Patients with histologically or pathologically confirmed non-Hodgkin lymphoma or malignant lymphoma, regardless of gender, 18 to 75 years of age (including the upper limit), are scheduled to undergo autologous hematopoietic stem cell transplantation; 3. Physical status of the Eastern Cancer Collaboration Group (ECOG) : the score was 0~2, and the expected survival time was more than 3 months; 4. Patients judged by researchers to be suitable for stem cell transplantation:

  1. Consolidation therapy after first-line induction chemotherapy for aggressive non-Hodgkin lymphoma with poor prognostic factors;
  2. It is suitable for salvage treatment of chemotherapy-sensitive non-Hodgkin lymphoma after recurrence;
  3. and salvage treatment of relapsed or primary refractory Hodgkin lymphoma that is sensitive to chemotherapy.

  5. The main organs function normally, the specific criteria are as follows:
  1. Bone marrow hematopoietic function is basically normal, blood routine: WBC ≥ 2.0×10^9/L, ANC ≥ 1.0×10^9/L, PLT ≥50×10^9/L, Hb ≥ 80 g/L. If the peripheral blood indexes were abnormal due to lymphoma invading bone marrow or spleen, the researchers could determine whether the patients were suitable for inclusion.
  2. Lung function: forced expiratory volume in one second (FEV1) ≥60%, carbon monoxide dispersion (DLCO) ≥50%;
  3. Liver function: total bilirubin, ALT and AST <2×ULN (upper limit of normal); AST and ALT≤3 times the upper limit of normal (ULN), total bilirubin (TBIL) ≤1.5×ULN (if there is liver invasion, AST and ALT≤5×ULN are allowed);
  4. Renal function: serum creatinine ≤1.5×ULN, creatinine clearance (CrCl) ≥ 60 ml/min (calculated according to Cockcroft-Gault formula). Male subjects: CLcr =[(140- age (years) x body weight (kg)) /[72 x serum creatinine (mg/dL)]; Female subjects: CLcr=0.85× CLcr of male subjects;
  5. Coagulation function: International standardized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5×ULN;
  6. Normal cardiac function: echocardiography or nuclide cardiac function test showed LVEF ≥ 55%, no uncontrolled tachycardia or Tachycardia syndrome, normal or abnormal ECG examination had no clinical significance, myocardial enzyme spectrum CK-MB was normal, pro-BNP was less than 900 pg/ml.

  6. Sufficient autologous hematopoietic stem cells have been assessed and collected by researchers: CD34≥2×106/Kg; 7. The women were not lactating, were not pregnant, and the female subjects with reproductive capacity were tested for serum pregnancy within 2 weeks before enrollment Test negative and agree not to become pregnant during the study period and for 36 months thereafter; Fertile male or female subjects must use a highly effective contraceptive method throughout the trial and for 1 year after the transplant.

Exclusion Criteria:

* 1. Received doxorubicin or anthracycline treatment in the past, and the total cumulative dose of doxorubicin was > 360 mg/m² (1 mg doxorubicin is equivalent to 2 mg epirubicin for other anthracycline drugs).

  2. Hypersensitivity to any investigational drug or its ingredients. 3. Cardiac function and disease consistent with one of the following conditions: a. Long QTc syndrome or QTc interval >480 ms; b. Complete left bundle branch block, degree II or III atrioventricular block; c. Severe, uncontrolled arrhythmias requiring medical treatment; d. New York College of Cardiology Grade ≥ III; e. Cardiac ejection fraction (LVEF) less than 50%; f. A history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities within the 6 months prior to recruitment.

  4. Hepatitis B, hepatitis C active infection (hepatitis B virus surface antigen or core antibody positive and hepatitis B virus DNA ultra Over 1×10³ copy /mL; More than 1×10³ copies /mL of HCV RNA). 5. Human immunodeficiency virus (HIV) infection (HIV antibody positive). 6. Previous or current co-occurrence of other malignancies (with the exception of malignancies with no known active disease occurring for ≥5 years prior to enrollment that have been treated for the purpose of cure); Basal cell carcinoma of the skin that has been adequately treated and shows no signs of disease (except melanoma); Well-treated carcinoma in situ of the cervix with no signs of disease).

  7. Have primary or secondary central nervous system (CNS) lymphoma or have a history of CNS lymphoma.

  8. Pregnant and lactating women and patients of childbearing age who do not want to take contraceptive measures.

  9. Patients who cannot collect CD34 + hematopoietic stem cells in quantities greater than or equal to 2×10^6/kg.

  10. Patients who have previously received solid organ transplants. 11. Patients who have received secondary or higher surgery within three weeks prior to treatment.

  12. Serious and active infectious diseases requiring systemic antibiotics, antifungal drugs, and antiviral treatment were present within 15 days prior to transplantation.

  13. People with a history of drug abuse (non-medical use of narcotic drugs or psychotropic drugs) or dependence on drugs (sedatives, hypnotics, analgesics, narcotics, stimulants and psychotropic drugs, etc.).

  14. Have a history of severe neurological or mental illness, including dementia or epilepsy.

  15. History of mental illness or cognitive impairment. 16. Patients deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lymphoma subjects for autologous hematopoietic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation | 100 days after transplantation
  Adverse reactions associated with pretreatment were evaluated in the United States in 2017. Published by the Department of Health and Human Services, see Glossary of Adverse Reactions Assessment (CTCAE5.0). Transplant-related mortality (TRM) was defined as treatment-related mortality not associated with the primary disease within 100 days of transplantation.

SECONDARY OUTCOMES:
Overall survival (OS) time | Time range: 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after transplant
  From transplant initiation to death or last follow-up
Progression-free survival (PFS) time | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after transplantation
  Time from the start of transplantation to disease progression, recurrence, death, or last follow-up

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Redondo AM, Valcarcel D, Gonzalez-Rodriguez AP, Suarez-Lledo M, Bello JL, Canales M, Gayoso J, Colorado M, Jarque I, Del Campo R, Arranz R, Terol MJ, Rifon JJ, Rodriguez MJ, Ramirez MJ, Castro N, Sanchez A, Lopez-Jimenez J, Montes-Moreno S, Briones J, Lopez A, Palomera L, Lopez-Guillermo A, Caballero D, Martin A; Grupo Espanol de Linfomas y Trasplante Autologo de Medula Osea (GELTAMO). Bendamustine as part of conditioning of autologous stem cell transplantation in patients with aggressive lymphoma: a phase 2 study from the GELTAMO group. Br J Haematol. 2019 Mar;184(5):797-807. doi: 10.1111/bjh.15713. Epub 2018 Dec 12. PMID 30548583
- [Background] Chen YB, Lane AA, Logan B, Zhu X, Akpek G, Aljurf M, Artz A, Bredeson CN, Cooke KR, Ho VT, Lazarus HM, Olsson R, Saber W, McCarthy P, Pasquini MC. Impact of conditioning regimen on outcomes for patients with lymphoma undergoing high-dose therapy with autologous hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2015 Jun;21(6):1046-1053. doi: 10.1016/j.bbmt.2015.02.005. Epub 2015 Feb 14. PMID 25687795
- [Background] El-Najjar I, Boumendil A, Luan JJ, Bouabdallah R, Thomson K, Mohty M, Colombat P, Biron P, Tilly H, Pfreundschuh M, Cordonnier C, Sureda A, Cahn JY, Vernant JP, Gribben J, Cook G, Haynes AP, Ferrant A, Finel H, Montoto S, Dreger P; Lymphoma Working Party of the European Group for Blood and Marrow Transplantation (EBMT). The impact of total body irradiation on the outcome of patients with follicular lymphoma treated with autologous stem-cell transplantation in the modern era: a retrospective study of the EBMT Lymphoma Working Party. Ann Oncol. 2014 Nov;25(11):2224-2229. doi: 10.1093/annonc/mdu440. Epub 2014 Sep 5. PMID 25193988
- [Background] Mills W, Chopra R, McMillan A, Pearce R, Linch DC, Goldstone AH. BEAM chemotherapy and autologous bone marrow transplantation for patients with relapsed or refractory non-Hodgkin's lymphoma. J Clin Oncol. 1995 Mar;13(3):588-95. doi: 10.1200/JCO.1995.13.3.588. PMID 7884420
- [Background] Isidori A, Clissa C, Loscocco F, Guiducci B, Barulli S, Malerba L, Gabucci E, Visani G. Advancement in high dose therapy and autologous stem cell rescue in lymphoma. World J Stem Cells. 2015 Aug 26;7(7):1039-46. doi: 10.4252/wjsc.v7.i7.1039. PMID 26328019
- [Background] Liu HW, Seftel MD, Rubinger M, Szwajcer D, Demers A, Nugent Z, Schroeder G, Butler JB, Cooke A. Total body irradiation compared with BEAM: Long-term outcomes of peripheral blood autologous stem cell transplantation for non-Hodgkin's lymphoma. Int J Radiat Oncol Biol Phys. 2010 Oct 1;78(2):513-20. doi: 10.1016/j.ijrobp.2009.08.024. Epub 2010 Feb 4. PMID 20137862
- [Background] Musso M, Scalone R, Marcacci G, Lanza F, Di Renzo N, Cascavilla N, Di Bartolomeo P, Crescimanno A, Perrone T, Pinto A. Fotemustine plus etoposide, cytarabine and melphalan (FEAM) as a new conditioning regimen for lymphoma patients undergoing auto-SCT: a multicenter feasibility study. Bone Marrow Transplant. 2010 Jul;45(7):1147-53. doi: 10.1038/bmt.2009.318. Epub 2009 Nov 9. PMID 19898504
- [Background] Gisselbrecht C, Glass B, Mounier N, Singh Gill D, Linch DC, Trneny M, Bosly A, Ketterer N, Shpilberg O, Hagberg H, Ma D, Briere J, Moskowitz CH, Schmitz N. Salvage regimens with autologous transplantation for relapsed large B-cell lymphoma in the rituximab era. J Clin Oncol. 2010 Sep 20;28(27):4184-90. doi: 10.1200/JCO.2010.28.1618. Epub 2010 Jul 26. PMID 20660832